CLINICAL TRIAL: NCT05720065
Title: Peripheral TMD Pain Mechanisms and the Effect by Botulinum Toxin A. A Randomized, Controlled, Double-blind Study
Brief Title: Peripheral TMD Pain Mechanisms and the Effect by Botulinum Toxin A
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Malin Ernberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022-05453-01
Record Dates: First submitted 2023-01-07; First posted 2023-02-09 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular Disorders; Botulinum Toxin A; Myalgia; Randomized; Clinical Trial; Pain; Gene; Neural Plasticity
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin (Active Comparator): Single bilateral injection into three standardized points of the masseter muscles and two of the anterior temporalis muscle. The total dose administered is 100 U (10 U/point) which is dissolved in 1 mL of isotonic saline. Thus, 0.1 ml of botulinum toxin solution is injected in each point.
  Interventions: Drug: Botulinum toxin type A
- Isotonic saline (Placebo Comparator): Single injection of 1 mL isotonic saline (0.9 mg/mL) into the same five points per side in a similar manner as for botulinum toxin.
  Interventions: Drug: Isotonic saline 0,9%

INTERVENTIONS:
Drug: Botulinum toxin type A — Randomized double-blind administration
  Other Names: Botox®️ (100 U, AbbVie AB, Solna, Sweden)
  Arms: Botulinum toxin
Drug: Isotonic saline 0,9% — Randomized double-blind administration
  Other Names: Natriumklorid Braun (0,9 mg/mL, B. Braun Medical AB, Danderyd, Sweden)
  Arms: Isotonic saline

SUMMARY:
The goal of this clinical trial is to investigate the effect of botulinum toxin on neurons' plasticity in the masseter muscle in humans with and without painful myogenous temporomandibular disorders (TMDM). The main questions it aims to answer are:

* does treatment with botulinum toxin alter gene expressions, epigenetic signatures, and cells plasticity in the masseter muscles of TMDM patients?
* do any such changes differ between patients with local and regional TMDM?
* does treatment with botulinum toxin influence pain characteristics (intensity, frequency, and sensibility) and other variables in patients with TMDM and are there correlations between significantly changed expression of biomarkers and other variables?

Participants will be examined with a questionnaire, clinical examination (including quantitative sensory testing; QST), and microbiopsy sampling from one of the masseter (MM) and anterior tibialis (AT) muscles and are then randomized to treatment with botulinum toxin or control (isotonic saline). Follow-ups occur after one and three months for all patients, and six months with questionnaire, clinical examination, and collection of post-treatment microbiopsies to see if botulinum toxin alter peripheral molecular events and clinical variables.

DETAILED DESCRIPTION:
Patient recruitment:

The patients will be recruited among those referred to the Specialist Clinic for Orofacial Pain and Jaw Function at the University Dental Clinic, Karolinska Institutet, Huddinge, Sweden, or via advertisement.

Randomization:

Patients will be randomly assigned to treatment by a random generator (www.randomization.com). For each participant the treatment will be written on a note and placed in a sealed envelope by a researcher not involved in any other part of data collection. A second person not involved in patient examination will open the envelope, prepare the syringe with the randomized solution, and place it in the examination room before the examiner and patient enters it. Botulinum toxin and saline have identical appearance so the participant and investigator will be masked to treatment assignment.

Procedure:

The participants complete an extended and slightly modified version of the Swedish Axis II questionnaire included in the Diagnostic Criteria for TMD (DC/TMD) before the first visit. The Axis II questionnaire contains sociodemographic question, questions regarding TMD symptoms and headache (presence, duration, and frequency) used for diagnostic purposes (Symptom Questionnaire), and validated instruments to assess physical and emotional function. A clinical examination is then performed according to the DC/TMD Axis I to ensure that the participant fulfils the enrollment criteria. If so, consent is signed. Then quantitative sensory testing (QST; thermal thresholds, pin-prick pain, temporal summation pain, pressure pain threshold, and conditioned pain modulation) is done and biopsies are obtained from a painful (MM) and a non-painful site (AT) for later analysis. At least one week hereafter treatment are given.

Axis II questionnaire:

For physical function the following instruments are used: PROMIS physical function short form (6b) to assess general physical function, the Oral Behavior Checklist (OBC) to assess presence and frequency of oral parafunctions, and the Jaw Functional Limitation Scale (JFLS).

To assess emotional function these instruments are included: The patient Health Questionnaire (PHQ-8) to screen for depression, the Generalized Anxiety Disorder (GAD-7), the Pain Catastrophizing Scale (PCS), the Perceived Stress Scale (PSS-10), the PROMIS sleep disturbance short form (6a) questionnaire, and the Oral Health Impact Profile (OHIP-5) to assess oral health-related quality of life.

Biopsies:

Microbiopsies will be obtained from one of the MA and the AT on the same side (a non-treated pain-free internal control). The microbiopsies are taken through the skin overlaying the most prominent part of the muscle under skin surface anesthesia. A disposable biopsy instrument with a penetration depth of 10 mm and a diameter of 18 gauche (G) (MM) or 16G (AT) are used. The biopsy instrument will be guided with a coaxial needle, that will be inserted to a depth of 10 mm. Maximum four microbiopsies are taken from each muscle to ensure that sufficient muscle tissue is obtained. The coaxial needle will be inserted along the long axis of the muscles until the fascia is penetrated and the biopsy instrument is then inserted through the coaxial needle and a piece of the muscle with a size of approximately 0.12 cm * 1.1 cm is collected. The muscle section will be removed from the biopsy instrument using a sterile probe and immediately put in a cryotube which is snap frozen in liquid nitrogen. After removal of the muscle section the biopsy instrument will be rinsed with isotonic saline. This procedure will be repeated three times (if possible). Each time the biopsy instrument will be rotated 45° so that the microbiopsy would be taken from a new portion of the muscle. The biopsies will be stored (-80º) in Karolinska Institutet's dental biobank until analysis.

Treatment:

Patients in the active treatment group receive 100 IU of botulinum toxin dissolved in 1 ml of isotonic saline. This dose is far below the lethal dose of 40 IU/kg body weight and is commonly used for treatment of TMD. In each MM 30 IU is injected divided between three different points (origin, mid-portion, and attachment) and in each temporalis muscle 20 IU (anterior and mid-inferior portion) after careful aspiration. Thus, in each point 10 IU of solution is injected. The solution is injected with EMG guidance using an audio-amplified device (Allergan Norden AB) to ensure intramuscular administration. A 1-mL syringe with a 19 mm needle (diameter 0.4 mm) will be used. Patients on the control treatment group receive intramuscular injection with isotonic saline (0.9%) in the same manner.

Analyses of biopsies:

The biopsies will be analyzed with bulk ribonucleic acid sequencing (RNA-seq) and single-cell seq including spatial transcriptomics at University of Texas Health Science Center in San Antonio (UTHSCSA). Flow cytometry (FC) analyses will be done at the ANA Futura lab in Huddinge, Sweden. IHC will be performed at the Live Cell Imaging Facility at Karolinska Institutet, Huddinge, Sweden, and proteomics at SciLife lab in Solna, Sweden. Data of the non-painful site (AT) will be subtracted from data of the painful site (MM) for every patient. Then, these data can be clustered.

For bulk RNA seq, differentially expressed genes (DEGs) will be selected and then paired analysis will be run within empirical analysis of DEGs in R (edgeR) software to select significantly different (p<0.05) DEGs. This is an established and well standardized approach. Selection criteria for further analysis are fold charge (FC)>1.5 and Reads Per Kilobase of transcript per Million mapped reads (RPKM)>10. Finally, biological processes will be defined by www.pantherdb.org on base of DEGs. Subtraction of internal controls from experimental data will also be done, followed by clustering of patients according to transcriptional profiles using K-mean principial component analysis algorithm. This last analysis is critical to build association of TMDM patient phenotypes with gene plasticity in MM and will be done with artificial intelligence (AI) and data learning (DL) algorithms by the Bioinformatics and Data Science Core (BDSC) at UTHSCSA. ScRNA-seq will be analyzed by SEURAT, which is by far more precise than standard clustering software from 10x Genomics.

The IHC analysis will focus on sensory neurite plasticity using markers for subsets of sensory neurons and use Light Sheet microscopy to measure neurite length and branching for whole biopsies. The following markers will primarily be used: PGP9.5, NFH, MrgprD, HTR3A, Nav 1.8, TrkA, TrkB, TrkC, MrgprA3, SP, CGRP, TRPV1, parvalbumin, calbindin, somatostatin, and PENK, but other markers can be considered as well. We also plan to use the Glyclick method which generates stable and homogenous antibody conjugates for IgG from several species and subclasses. FC will be used to profile immune and vasculature cells.

Proteomics will be done with two methods. First two-dimensional gel electrophoresis followed by identification with liquid chromatography-tandem mass spectrometry, followed by protein network analyses. Therafter affinity proteomics using Olink platforms will be done, which enables analysis of several hundreds of proteins in one analysis.

When all the analyses are done and the results published any remaining material will be discarded.

When the analyses at UTHSC are done, and the results published any remaining material will be discarded. If any material is remaining from samples in Sweden, they will be kept in the dental biobank at KI for other analyses.

Statistical analyses of primary outcomes (biological markers):

Pilot experiments show that 20 patients in each group are needed to attain >80% power for each test detecting at least 2-fold significant difference (FC) in gene expression with an estimated standard deviation of 0.6 (considering high human-to-human variation; this includes samples after botulinum toxin treatment. Power analysis show that we need 10 paired samples per group for scRNA seq, IHC and FC. To obtain sufficient power data from 40 patients will be included in proteomic analyses, which will give a power of 0.856 with an expected difference from baseline at the 1-mo follow-up of 20% (SD 30%) with alpha = 0.050 and beta = 0.20 (paired t-test).

Statistical analyses will be done with 1-, 2- and 3-way and repeated measures ANOVA with Bonferroni's post-hoc test. For scRNA seq, currently accepted analysis for is that paired samples belonging to the same participant group combined and multiple t-test-like analysis for each cell cluster run against another group. Prism v8 software (GraphPad Software LLT, Boston, MA, USA) will be used with p < 0.05 as significance level.

Statistical analyses of secondary outcomes (clinical data):

Even if the sample size is not calculated based on clinical data, power analysis for pain intensity based on a previous study show that 20 patients per arm would yield a power of 0.977 given a group difference of 3.14 (SD 2.45) and a significance level of p < 0.05. Given the invasive nature of the project (repeated microbiopsies) a relatively high drop-out rate is expected why 5 additional participants will be recruited per group (MYA, MFP, healthy controls).

For statistical univariate analyses the SigmaPlot v 14 software will be used (Systat Software Inc, Chicago, IL, USA). Mean (SD) or median (interquartile range, IQR), depending on normality, will be used to describe the data. To compare groups in Project A, ANOVA or Kruskall-Wallis' test will be used. Repeated measures ANOVA with Dunnet's posthoc test will be used the analyze differences in treatment effect with Group and time as factors in Project B. Data that are skewed or ordinal (most Axis II data) will be analyzed with Friedman ANOVA for each group separately with Dunn's test as posthoc test for time differences. The Mann-Whitney U-test will be used to analyze differences between groups at different time points, using Bonferroni correction for multiple testing. Differences are considered as significant when p < 0.05.

Further, multivariate statistics will be used to identify correlations between significantly changed biomarkers and other variables using SIMCA v.17.0 (Sartorius Stedim Biotech, Umeå, Sweden). Principal component analysis (PCA) will be used to identify moderate or strong outliers. Orthogonal partial least squares discriminant analysis (OPLS-DA) will then be used to regress group membership using the biomarkers as regressors. For correlations between biomarkers and clinical variables OPLS modeling will be performed. The variable in-fluence on projection (VIP) value indicates the relevance of each X-variable pooled over all dimensions and the Y-variables indicate the group of variables that best explain Y. VIP > 1.0 is considered significant. R2 describes the goodness of fit, i.e., the fraction of sum of squares of all the variables explained by a principal component whereas Q2 describes the goodness of prediction, i.e., the fraction of the total variation of the variables that can be predicted by a principal component using cross validation methods. R2 should not be considerably higher than Q2, if substantially higher (>0.3) the robustness of the model is poor. To validate the model, an obtained CV-ANOVA p-value will be used. The OPLS-DA model is considered of significant importance if the CV-ANOVA has a p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of TMDM myalgia or myofascial pain according to the DC/TMD criteria
* females with adequate contraceptives and a negative pregnancy test
* pain upon digital palpation of at least one of the masseter muscle
* a characteristic pain intensity of > 40/100
* a negative pregnancy test at the day of treatment

Exclusion Criteria:

* difficulties understanding the Swedish language
* systemic inflammatory connective tissue diseases
* widespread pain
* neuromuscular disorders
* diagnosed or severe psychiatric disease
* neuropathic pain
* pain of dental origin
* history of trauma to the face, head or neck
* pregnancy or nursing
* known allergy to botulinum toxin or antibiotics
* use of muscle relaxants, antidepressant, neuropsychiatric, anticoagulant drugs, or aminoglycoside antibiotics
* previous treatment with botulinum toxin during the last 12 months
* use of analgesic or anti-inflammatory medication during the 48 hours preceding biopsy
* skin infection over injection/biopsy site

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of gene expression measured with bulk RNA-seq | 1-6 months
  Gene expression in the anterior tibialis muscle (internal control) will be subtracted from the masseter and the patients will then be clustered according to DEGs and compared to baseline.
Change of RNA expression measured with single-cell RNA (scRNA) seq/spatial trnascriptomics. | 1-6 months
  ScRNA-seq will be analyzed by SEURAT
Change of expression of sensory neuron markers measured with IHC | 1-6 months
  The expression will be measured as the change of frequency (%) of selected sensory neuron markers.
Change of proteome measured with proteomics | 1-6 months
  The expression wil be measured with two-dimensional gel electrophoresis, followed by liquid chromatography-tandem mass spectrometry and protein network analyses.
Change of proteome measured with affinity-based proteomics. | 1-6 months
  The protein expression will be measured with affinity proteomics using Olink platforms will be done, which enables analysis of several hundreds of proteins in one analysis

SECONDARY OUTCOMES:
Change of pain intensity compared to baseline using 0-10 numeric rating scales (NRS) | 1-3 months
  Assessed with the Brief Pain Inventory and includes assessment of the current and the worst, average, and least pain intensity during the last week, each scored on 0-10 numeric rating scale. The worst, average, and current pain can be used to calculate the Characteristic Pain Intensity (0-100) which is the mean score of the three assessments multiplied with ten.
Global improvement using Patient Global Impression of Change Scale (PGIC) | 1-3 months
  Assessed with the 7-point PGIC with the alternatives: 0 = eliminated, 1 = much improved, 2 = improved, 3 = unchanged, 4 = impaired, 5 =much impaired and 6 = very much impaired.
Change of pain quality compared to baseline using the McGill Pain questionnaire (MPQ) | 1-3 months
  Assessed with the MPQ Short-Form which includes 15 adjectives that can be used to describe pain, each scored according to severity (0-3). The total score is calculated.
Number of participants with adverse events assessed with questionnaire | 1 week
  The participant lists any adverse event occurring during the week after injection and rate them as mild, moderate or severe.
Number of participants with adverse events assessed with questionnaire | 1-3 months
  The participant lists any adverse event occurring since the last visit and rate them as mild, moderate or severe.
Change of physical function assessed with questionnaire | 1-3 months
  Assessed with the Axis II questionnaire included in the DC/TMD. Includes the The Brief Pain Inventory (7 items, score ranges 0-100 for each), the Jaw Function Limitation Scale (20 items, score ranges 0-10), and the Oral Behavior Checklist (21 items, score ranges 0-84). A lower score indicates a better outcome for all instruments.
Change of emotional function assessed with questionnaire | 1-3 months
  Assessed with the Axis II questionnaire included in the DC/TMD. Includes the Beck's Depression inventory (21 items, score ranges 0-63), the Generalized Anxiety Disorder (7 items, score ranges 0-21), the Patient Health Questionnaire (15 items, score ranges 0-30), the Pain Catastrophizing Scale (13 items, score ranges 0-52), the Perceived Stress Scale (1o items, score ranges 0-40), and the Insomnia Severity Index (7 items, score ranges 0-28). A lower score indicates a better outcome for all instruments.

OTHER OUTCOMES:
Change of thermal detection and pain thresholds measured with Thermotest. | 1-3 months
  The program is set at first recording warmth (WST) and cold detection thresholds (CDT) four times and then cold (CPT) and heat pain thresholds (HPT) three times. The mean of the recording for each threshold is calculated by the program software and used in analyses.
Change of pin-prick pain measured with Medipin | 1-3 months
  The perceived magnitude of a single pin-prick stimulus is assessed using a Medipin® (Medipin Limited, Hertfordshire, United Kingdom). The device is applied perpendicular to the skin for 1-2 seconds. Then the participant is asked to give a pain rating representing the pain at the end of the stimuli using a 0-100 NRS.
Change of temporal summation pain compared to baseline | 1-3 months
  Temporal summation will be evoked with a 1.0 kg palpometer. The stimulus will be applied 10 times at the masseter muscle for 2 s with 1 s interval and pain intensity will be recorded after the 1st, 5th, and 10th stimulation on a 0-10 NRS.
Change of pressure pain threshold (PPT) compared to baseline | 1-3 months
  The PPT (kPa) will be recorded over the masseter muscle with an electronic algometer as the average of three recordings
Change of conditioned pain modulation (CPM) compared to baseline | 1-3 months
  During CPM the participant immerse her hand and wrist into a cold water bath during 60s. The PPT (kPa) is recorded immediately before and after hand immersion. The percent change (%) before-after is used as CPM value.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Ernberg, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Dental Medicine, Karolinska Institutet, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Deidentified genetic and other data will be entered into a database at the National Institute of Health (NIH) that only contains genetic data, sex, age, and TMD diagnosis.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be available after study termination and saved in the databases for 10 years whereafter they are discarded.
Access Criteria: The database is made available to other researchers only for non-commercial research that has permission from the ethics committee after approval by the research leader (controlled access). Data is also uploaded into a database of aggregated genomic data that is shared with the research community (unlimited access).

REFERENCES:
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Ernberg M, Hedenberg-Magnusson B, List T, Svensson P. Efficacy of botulinum toxin type A for treatment of persistent myofascial TMD pain: a randomized, controlled, double-blind multicenter study. Pain. 2011 Sep;152(9):1988-1996. doi: 10.1016/j.pain.2011.03.036. Epub 2011 Apr 22. PMID 21514731
- [Background] Mecklenburg J, Wangzhou A, Hovhannisyan AH, Barba-Escobedo P, Shein SA, Zou Y, Weldon K, Lai Z, Goffin V, Dussor G, Tumanov AV, Price TJ, Akopian AN. Sex-dependent pain trajectories induced by prolactin require an inflammatory response for pain resolution. Brain Behav Immun. 2022 Mar;101:246-263. doi: 10.1016/j.bbi.2022.01.016. Epub 2022 Jan 19. PMID 35065194
- [Background] Srzentic K, Fornelli L, Tsybin YO, Loo JA, Seckler H, Agar JN, Anderson LC, Bai DL, Beck A, Brodbelt JS, van der Burgt YEM, Chamot-Rooke J, Chatterjee S, Chen Y, Clarke DJ, Danis PO, Diedrich JK, D'Ippolito RA, Dupre M, Gasilova N, Ge Y, Goo YA, Goodlett DR, Greer S, Haselmann KF, He L, Hendrickson CL, Hinkle JD, Holt MV, Hughes S, Hunt DF, Kelleher NL, Kozhinov AN, Lin Z, Malosse C, Marshall AG, Menin L, Millikin RJ, Nagornov KO, Nicolardi S, Pasa-Tolic L, Pengelley S, Quebbemann NR, Resemann A, Sandoval W, Sarin R, Schmitt ND, Shabanowitz J, Shaw JB, Shortreed MR, Smith LM, Sobott F, Suckau D, Toby T, Weisbrod CR, Wildburger NC, Yates JR 3rd, Yoon SH, Young NL, Zhou M. Interlaboratory Study for Characterizing Monoclonal Antibodies by Top-Down and Middle-Down Mass Spectrometry. J Am Soc Mass Spectrom. 2020 Sep 2;31(9):1783-1802. doi: 10.1021/jasms.0c00036. Epub 2020 Aug 19. PMID 32812765
- [Background] Christidis N, Kang I, Cairns BE, Kumar U, Dong X, Rosen A, Kopp S, Ernberg M. Expression of 5-HT3 receptors and TTX resistant sodium channels (Na(V)1.8) on muscle nerve fibers in pain-free humans and patients with chronic myofascial temporomandibular disorders. J Headache Pain. 2014 Sep 26;15(1):63. doi: 10.1186/1129-2377-15-63. PMID 25261281
- [Background] Wheelock AM, Wheelock CE. Trials and tribulations of 'omics data analysis: assessing quality of SIMCA-based multivariate models using examples from pulmonary medicine. Mol Biosyst. 2013 Nov;9(11):2589-96. doi: 10.1039/c3mb70194h. PMID 23999822
- [Background] De la Torre Canales G, Alvarez-Pinzon N, Munoz-Lora VRM, Vieira Peroni L, Farias Gomes A, Sanchez-Ayala A, Haiter-Neto F, Manfredini D, Rizzatti-Barbosa CM. Efficacy and Safety of Botulinum Toxin Type A on Persistent Myofascial Pain: A Randomized Clinical Trial. Toxins (Basel). 2020 Jun 15;12(6):395. doi: 10.3390/toxins12060395. PMID 32549196
- See also: Random generator — http://www.jerrydallal.com/random/randomize.htm